CLINICAL TRIAL: NCT07059156
Title: Multicenter Study on Integrated Treatment Regimen of Induction-Consolidation Chemotherapy and Transplantation for Adult Acute Lymphoblastic Leukemia
Brief Title: Multicenter Study of Combined Chemotherapy and Transplantation for Adult ALL
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShanxiBethuneH1
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphoblastic Leukemia, Adult
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multicenter Study of Combined Chemotherapy and Transplantation for Adult ALL (Experimental)
  Interventions: Drug: Induction Therapy Regimen; Drug: Pre-Treatment Regimen; Other: Post-CR Treatment; Drug: Post-CR Consolidation Regimens; Other: Transplant-Eligible Subsequent Therapy; Other: Allo-HSCT Protocol; Other: Non-Transplant Maintenance Therapy Options

INTERVENTIONS:
Drug: Induction Therapy Regimen — VICP+VEN regimen:
  * Vindesine: 3 mg/m²/day (max 4 mg), administered on days 1, 8, 15, 22.
  * Idarubicin (IDA): 8 mg/m², days 1, 8, 15, 22.
  * Cyclophosphamide (CTX): 500 mg/m², days 7, 21.
  * Prednisone: 1 mg/kg/day, days 1-14; 0.5 mg/kg/day, days 15-28
  * Venetoclax (VEN) 8-day ramp-up: Day 1: 100 mg, Day 2: 200 mg, Days 3-8: 400 mg/day
Drug: Pre-Treatment Regimen — Indications for pre-treatment:
  * WBC ≥30×10⁹/L, or significant hepatosplenomegaly/lymphadenopathy.
  * Laboratory signs of tumor lysis syndrome (e.g., electrolyte abnormalities).
  Pre-treatment protocol:
  * Glucocorticoids (e.g., prednisone or dexamethasone): Prednisone 1 mg/kg/day (PO/IV) for 3-5 days.
  * Optional addition of CTX: 200 mg/m²/day IV for 3-5 days.
Other: Post-CR Treatment — Principles:
  1. MRD-positive or rising: Administer blinatumomab (CD19/CD3 bispecific antibody) for residual disease clearance, followed by allogeneic hematopoietic stem cell transplantation (allo-HSCT).
  2. MRD-negative/unknown: Continue multi-agent chemotherapy ± blinatumomab consolidation. Allo-HSCT for patients with high-risk clinical/genetic features.
Drug: Post-CR Consolidation Regimens — ① Hyper-CVAD-B (Methotrexate/Cytarabine-based):
  * Methotrexate (MTX): 1 g/m² IV over 24h (Day 1) with urine alkalinization (pH >7.0) and leucovorin rescue.
  * Cytarabine (Ara-C): 1 g/m² IV q12h (Days 2-3; total 4 doses).
  * Dexamethasone: 40 mg/day (PO/IV, Days 1-4).
  * Cycle interval: 21-28 days (alternating with other regimens).
    ② CAM Regimen:
  * CTX: 750 mg/m² IV (split over 2 days).
  * Ara-C: 75 mg/m²/dose (8 days; 1-2 doses/day IV; if once daily, administer 5 days/week × 2 weeks).
  * 6-MP: 50-75 mg/m²/day fasting (7-14 days PO).
Other: Transplant-Eligible Subsequent Therapy — * Allo-HSCT for eligible patients after induction.
  * Conditioning regimen: TBI-VP16-CY.
  * Donor priority: HLA-matched sibling donor (MSD), Matched unrelated donor (MUD), Haploidentical donor (Haplo).(Consider age/donor health status).
Other: Allo-HSCT Protocol — 1.6.1 Conditioning Regimen (TBI-VP16-Cy/ATG):
  * TBI: 5 Gy (Days -7 to -6).
  * VP16: 10 mg/kg/day (Days -5 to -4).
  * CTX: 30 mg/kg/day (Days -3 to -2).
  * ATG: 7.5 mg/kg/day (Days -5 to -2). 1.6.2 GVHD Prophylaxis:
  * Basiliximab (anti-CD25 mAb): 50 mg (Days +1, +4).
  * Standard regimen: Cyclosporine (CsA): IV: 2 mg/kg/day (start Day -9; target level 150-250 μg/L). PO: 3-5 mg/kg/day BID (switch delayed until Day +10 if no aGVHD); Mycophenolate mofetil (MMF) + short-course methotrexate.
Other: Non-Transplant Maintenance Therapy Options — ① Hyper-CVAD-B (Methotrexate/Cytarabine-based):
  * Methotrexate (MTX): 1 g/m² IV over 24h (Day 1) with urine alkalinization (pH >7.0) and leucovorin rescue.
  * Cytarabine (Ara-C): 1 g/m² IV q12h (Days 2-3; total 4 doses).
  * Dexamethasone: 40 mg/day (PO/IV, Days 1-4).
  * Cycle interval: 21-28 days (alternating with other regimens).
    ② CAM Regimen:
  * CTX: 750 mg/m² IV (split over 2 days).
  * Ara-C: 75 mg/m²/dose (8 days; 1-2 doses/day IV; if once daily, administer 5 days/week × 2 weeks).
  * 6-MP: 50-75 mg/m²/day fasting (7-14 days PO).
    * Maintenance (6-MP/MTX alternating with V-Dex): 6-MP: 75 mg/m²/day at bedtime (Days 1-21); MTX: 20 mg/m² IM weekly × 3 weeks.*Adjust doses to maintain WBC ~3×10⁹/L, ANC 1.0-1.5×10⁹/L.*

SUMMARY:
This study aims to evaluate an integrated treatment protocol for adults with Philadelphia chromosome-negative acute lymphoblastic leukemia (Ph- ALL), combining induction chemotherapy, consolidation therapy, and allogeneic hematopoietic stem cell transplantation (allo-HSCT) to improve treatment efficacy and survival rates. The single-arm, open-label, multicenter study will enroll 50 newly diagnosed patients aged 18-60 years. The induction phase employs the VICP+VEN regimen (vindesine, idarubicin, cyclophosphamide, prednisone combined with venetoclax), followed by consolidation therapy with either Hyper-CVAD or CAM protocols, with eligible patients proceeding to allo-HSCT. Primary endpoints include disease-free survival (DFS) and complete remission (CR) rates, while secondary endpoints encompass relapse rate, overall survival (OS), and safety. Patients will be followed for 2 years with regular monitoring of minimal residual disease (MRD) and adverse events. The protocol is designed to reduce relapse risk through intensive therapy and transplantation, offering a potential cure for high-risk patients.The goal is to complete the entire treatment within 4 months after diagnosis.

DETAILED DESCRIPTION:
1. Intervention Measures 1.1 Induction Therapy Regimen

VICP+VEN regimen:

* Vindesine: 3 mg/m²/day (max 4 mg), administered on days 1, 8, 15, 22.
* Idarubicin (IDA): 8 mg/m², days 1, 8, 15, 22.
* Cyclophosphamide (CTX): 500 mg/m², days 7, 21.
* Prednisone: 1 mg/kg/day, days 1-14; 0.5 mg/kg/day, days 15-28
* Venetoclax (VEN) 8-day ramp-up: Day 1: 100 mg, Day 2: 200 mg, Days 3-8: 400 mg/day 1.2 Pre-Treatment Regimen

Indications for pre-treatment:

* WBC ≥30×10⁹/L, or significant hepatosplenomegaly/lymphadenopathy.
* Laboratory signs of tumor lysis syndrome (e.g., electrolyte abnormalities).

Pre-treatment protocol:

* Glucocorticoids (e.g., prednisone or dexamethasone): Prednisone 1 mg/kg/day (PO/IV) for 3-5 days.
* Optional addition of CTX: 200 mg/m²/day IV for 3-5 days. 1.3 Post-CR Treatment

Principles:

1. MRD-positive or rising: Administer blinatumomab (CD19/CD3 bispecific antibody) for residual disease clearance, followed by allogeneic hematopoietic stem cell transplantation (allo-HSCT).
2. MRD-negative/unknown: Continue multi-agent chemotherapy ± blinatumomab consolidation. Allo-HSCT for patients with high-risk clinical/genetic features.

   1.4 Post-CR Consolidation Regimens

   ① Hyper-CVAD-B (Methotrexate/Cytarabine-based):
   * Methotrexate (MTX): 1 g/m² IV over 24h (Day 1) with urine alkalinization (pH >7.0) and leucovorin rescue.
   * Cytarabine (Ara-C): 1 g/m² IV q12h (Days 2-3; total 4 doses).
   * Dexamethasone: 40 mg/day (PO/IV, Days 1-4).
   * Cycle interval: 21-28 days (alternating with other regimens).

     * CAM Regimen:
   * CTX: 750 mg/m² IV (split over 2 days).
   * Ara-C: 75 mg/m²/dose (8 days; 1-2 doses/day IV; if once daily, administer 5 days/week × 2 weeks).
   * 6-MP: 50-75 mg/m²/day fasting (7-14 days PO). 1.5 Transplant-Eligible Subsequent Therapy
   * Allo-HSCT for eligible patients after induction.
   * Conditioning regimen: TBI-VP16-CY.
   * Donor priority: HLA-matched sibling donor (MSD), Matched unrelated donor (MUD), Haploidentical donor (Haplo). (Consider age/donor health status).

   1.6 Allo-HSCT Protocol 1.6.1 Conditioning Regimen (TBI-VP16-Cy/ATG):

   • TBI: 5 Gy (Days -7 to -6).
   * VP16: 10 mg/kg/day (Days -5 to -4).
   * CTX: 30 mg/kg/day (Days -3 to -2).
   * ATG: 7.5 mg/kg/day (Days -5 to -2). 1.6.2 GVHD Prophylaxis:
   * Basiliximab (anti-CD25 mAb): 50 mg (Days +1, +4).
   * Standard regimen: Cyclosporine (CsA): IV: 2 mg/kg/day (start Day -9; target level 150-250 μg/L). PO: 3-5 mg/kg/day BID (switch delayed until Day +10 if no aGVHD); Mycophenolate mofetil (MMF) + short-course methotrexate.

   1.7 Non-Transplant Maintenance Therapy

   Options:
   * Hyper-CVAD-B (Methotrexate/Cytarabine-based):

     • Methotrexate (MTX): 1 g/m² IV over 24h (Day 1) with urine alkalinization (pH >7.0) and leucovorin rescue.

     • Cytarabine (Ara-C): 1 g/m² IV q12h (Days 2-3; total 4 doses).

     • Dexamethasone: 40 mg/day (PO/IV, Days 1-4).
     * Cycle interval: 21-28 days (alternating with other regimens).

       * CAM Regimen:
     * CTX: 750 mg/m² IV (split over 2 days).
     * Ara-C: 75 mg/m²/dose (8 days; 1-2 doses/day IV; if once daily, administer 5 days/week × 2 weeks).
     * 6-MP: 50-75 mg/m²/day fasting (7-14 days PO).

       * Maintenance (6-MP/MTX alternating with V-Dex): 6-MP: 75 mg/m²/day at bedtime (Days 1-21); MTX: 20 mg/m² IM weekly × 3 weeks.*Adjust doses to maintain WBC ~3×10⁹/L, ANC 1.0-1.5×10⁹/L.*

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 60 years；
2. Diagnosis must comply with the Chinese Guidelines for Diagnosis and Treatment of Adult Acute Lymphoblastic Leukemia (2024 Edition), requiring MICM (Morphology, Immunology, Cytogenetics, and Molecular genetics) integration and WHO 2022 (5th edition) classification standards. The minimal diagnostic workup must include morphological assessment and immunophenotyping to differentiate ALL from acute myeloid leukemia (AML). All patients shall undergo bone marrow aspiration plus biopsy at initial diagnosis. A definitive ALL diagnosis requires ≥20% blasts/immature lymphocytes in bone marrow (Note: Patients with <20% blasts due to fever or glucocorticoid pretreatment require comprehensive evaluation incorporating medical history and ancillary tests for differential diagnosis)；
3. ECOG Performance Status: 0-2

Exclusion Criteria:

1. Intracranial hemorrhage
2. Pregnancy
3. Psychiatric disorders or other conditions compromising protocol compliance
4. Severe cardiac arrhythmia with ECG abnormalities (QTc >500 ms)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival (DFS) | 24 months
Complete remission (CR) rate | 24 months
Partial remission (PR) rate | 24 months
Non-remission (NR) rate | 24 months
CR with incomplete hematologic recovery (CRi) | 24 months

SECONDARY OUTCOMES:
Relapse rate | 24 months
Treatment-related mortality（TRM） | 24 months
Overall Survival（OS） | 24 months
Event-Free Survival（EFS） | 24 months
Adverse Event | 24 months
Mortality | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China